CLINICAL TRIAL: NCT06208137
Title: Using the Composite Immune Risk Score to Assess and Modulate the Patient's Immune Reconstitution After Allogeneic Hematopoietic Stem Cell Transplantation, a Prospective, Multicenter, Randomized Controlled Study.
Brief Title: Using the Composite Immune Risk Score to Assess and Modulate the Patient's Post-transplant Immune Reconstitution.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2023022
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-03

CONDITIONS: Transplant-Related Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Remind patients to test their immune status among 120-180 days post-transplantation. Physicians assessed the risk level of patients in the intervention group based on their immune status on days 91-180 using the CIRS.
  Interventions: Behavioral: Health monitoring and regular return follow-up reminders
- Control group (No Intervention): Only remind patients to test their immune status among 120-180 days post-transplantation.

INTERVENTIONS:
Behavioral: Health monitoring and regular return follow-up reminders — Health monitoring & reminders for blood tests and follow-up visits until 1 year post-transplant
  Arms: Intervention group

SUMMARY:
To assess the effectiveness of interventions including health monitoring and regular return follow-up reminders for patients with a high Composite Immune Risk Score.

DETAILED DESCRIPTION:
This study aims to prospectively evaluate the effectiveness of the Composite Immune Risk Score in real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients must be ≥ 16 years of age;
* 2) Patients receiving haploidentical allo-HSCT;
* 3) Patients have to sign an informed consent form before the start of the research procedure.

Exclusion Criteria:

* 1) Tandem transplantation or multiple transplantations;
* 2) Mental or other medical conditions that make the patients unable to comply with the research treatment and monitoring requirements;
* 3) Patients who are ineligible for the study due to other factors, or will bear great risk if participating in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 1.5 years after transplantation
  Overall survival during 1.5 years after transplantation

SECONDARY OUTCOMES:
Non-relapse mortality rate | 1.5 years after transplantation
  Non-relapse mortality rate during 1.5 years after transplantation
Incidence of infections | 1.5 years after transplantation
  Infections during 1.5 years after transplantation
Immune cell count | 1.5 years after transplantation
  Data on immune cell count will be collected during 1.5 years after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT06208137/Prot_001.pdf